CLINICAL TRIAL: NCT02079597
Title: Prospective Study to Analyze Ninjurin-1 and Its Soluble Part During Systemic Inflammation
Brief Title: The Role of Ninjurin-1 During Systemic Inflammation
Acronym: Ninj1
Status: Completed | Type: Observational
Sponsor: Dr. Patrick Meybohm, M.D. (Other)
Responsible Party: Sponsor-Investigator, Dr. Patrick Meybohm, M.D., PD Dr. Patrick Meybohm, M.D., Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Other Study IDs: NINJ1-001
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Ninj1 Expression; SIRS
Keywords: SIRS; Ninj1; Sepsis; Healthy
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma, RNA and cDNA extracted from whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy: Healthy individuals no infection
- SIRS: SIRS patients no included in an interventional study no peroperative infection

SUMMARY:
* With the underlying study the investigators address the question if Ninjurin-1 (Ninj1) expression is altered in patients with systemic inflammatory response syndrome (SIRS) in comparison to healthy volunteers.
* The adhesion molecule Ninj1 is induced following nerve injury where it contributes to nerve generation. Besides it is described to facilitate leukocyte migration especially in the nervous system.
* The investigators hypothesize that Ninj1 expression is increased in SIRS patients, which will fortify its impact during inflammation and the transferability from bench to bedside.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* cardiac surgery patients

Exclusion Criteria:

* included in an interventional study
* Preoperative Infection (e.g. Endocarditis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SIRS patients: Intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Ninj1 expression on blood leukocytes | one day post surgery

SECONDARY OUTCOMES:
grade of systemic inflammation | one day post surgery
  routine inflammatory markers will be used to evaluate the grade of inflammation e.g. procalcitonin (PCT) Interleukin 6, lipopolysaccharide (LPS) binding protein (LBP). Retrospective evaluation for sepsis (bacterial infection)

OTHER OUTCOMES:
Soluble Ninj1 concentration/expression rates | one day post surgery
  Concentration will be measured in plasma samples as well as from whole blood culture incubated with 100 ng/ml lipopolysaccharide for 6, 16 and 24 h.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meybohm, MD, Principal Investigator — Department of Anesthesiology, University Hospital Frankfurt
Locations (1):
- Department of Anesthesiology, University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany